CLINICAL TRIAL: NCT07248774
Title: Effect of Bubble Positive Expiratory Pressure and Segmental Breathing Versus Incentive Spirometry on Lung Expansion and Dyspnea in Children With Pleural Effusion
Brief Title: Effect of Bubble Positive Expiratory Pressure and Segmental Breathing Versus Incentive Spirometry in Pleural Effusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/TAYYBABARI
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pleural Effusion
Keywords: Pleural effusion, PEP, Segmental Breathing, Dyspnea
MeSH Terms: conditions — Pleural Effusion; Dyspnea

STUDY DESIGN:
Intervention Model Description: Conducted as a randomized clinical trial, this study will include 40 pediatric participants aged 5-16, recruited from Gulab Devi Chest Hospital and Children's Hospital, Lahore. Participants will be randomly divided into two groups: one receiving Bubble PEP with Segmental Breathing and the other using Incentive Spirometry, both combined with conventional chest physiotherapy and mobility. Outcome measures, including lung expansion (via X-ray), dyspnea (assessed using the Pediatric Dyspnea Scale), chest expansion (measured with a measuring tape), oxygen saturation (SpO₂), and respiratory rate, will be recorded pre- and post-intervention. The study hypothesises that the Bubble PEP and Segmental Breathing approach may offer a cost-effective and efficient alternative to Incentive Spirometry, particularly for patients who cannot afford mechanical devices. Statistical analysis will be performed using SPSS version 2023 to determine the intervention's effects.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols, and possible efforts will be put to mask both groups about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Intervention Group (Bubble PEP + Segmental Breathing) (Active Comparator): The experimental group will receive Bubble PEP therapy and Segmental Breathing along with conventional chest physiotherapy and mobility training. Bubble PEP will be performed using a bottle device where children exhale through a water-submerged tube, creating resistance to improve lung expansion and secretion clearance (10 repetitions, progressing from 1 to 3 sets over 14 days). Segmental Breathing will focus on localized lung expansion with therapist-guided tactile feedback, performed at six breaths per minute, progressing from 1 to 3 sets. Chest percussion will be applied for 2-5 minutes with rest intervals, and walking distance will increase from 1 to 5 meters. All sessions will be conducted once daily for two weeks.
  Interventions: Other: Bubble PEP
- Group B: Control Group (Incentive Spirometry) (Active Comparator): Participants in the control group will receive Incentive Spirometry along with conventional chest physiotherapy and mobility training. Incentive Spirometry will be used to encourage sustained maximal inspiration, thereby promoting lung expansion and improving ventilation. Each session will include three repetitions per side during Days 1-3, five repetitions per side during Days 4-7, and ten repetitions per side during Days 8-14, performed in one set per session. Chest percussion will be administered on the contralateral side to facilitate secretion mobilization, performed for two minutes on Days 1-3, three minutes on Days 4-7, and five minutes on Days 8-14, with 15 seconds of rest after each minute. Mobility training will include walking exercises, starting from one meter on Day 1, increasing to three meters by Day 3, and progressing to five meters from Day 4 onward, performed in two sets during Days 8-14. All sessions will be conducted once daily for two weeks.
  Interventions: Other: Incentive Spirometery

INTERVENTIONS:
Other: Bubble PEP — Bubble PEP will be performed using a bottle device with 10 repetitions, progressing from one to three sets over 14 days. Segmental Breathing will target localized lung expansion with six breaths per minute, progressing similarly. Chest percussion will be applied on the contralateral side for 2-5 minutes with rest intervals, and walking distance will increase from 1 to 5 meters across the intervention period. All sessions will be conducted once daily for two weeks, with pre- and post-intervention assessments of lung expansion and dyspnea.
  Other Names: Segmental Breathing
  Arms: Group A: Intervention Group (Bubble PEP + Segmental Breathing)
Other: Incentive Spirometery — Incentive Spirometry will be used to encourage sustained maximal inspiration, thereby promoting lung expansion and improving ventilation. Each session will include three repetitions per side during Days 1-3, five repetitions per side during Days 4-7, and ten repetitions per side during Days 8-14, performed in one set per session.
  Arms: Group B: Control Group (Incentive Spirometry)

SUMMARY:
Conducted as a randomized clinical trial, this study will include 40 pediatric participants aged 5-16, recruited from Gulab Devi Chest Hospital and Children's Hospital, Lahore. Participants will be randomly divided into two groups: one receiving Bubble PEP with Segmental Breathing and the other using Incentive Spirometry, both combined with conventional chest physiotherapy and mobility. Outcome measures, including lung expansion (via X-ray), dyspnea (assessed using the Pediatric Dyspnea Scale), chest expansion (measured with a measuring tape), oxygen saturation (SpO₂), and respiratory rate, will be recorded pre- and post-intervention. The study hypothesises that the Bubble PEP and Segmental Breathing approach may offer a cost-effective and efficient alternative to Incentive Spirometry, particularly for patients who cannot afford mechanical devices. Statistical analysis will be performed using SPSS version 2023 to determine the intervention's effects.

DETAILED DESCRIPTION:
Pleural effusion is the pathological accumulation of excess fluid in the pleural cavity, compromising lung function by limiting expansion and reducing compliance. This condition leads to symptoms such as dyspnea and impaired gas exchange, which can significantly affect pediatric patients. Treatment often includes physical therapy techniques to facilitate lung expansion and improve respiratory function. The present study comprises Bubble Positive Expiratory Pressure, which involves exhalation through water to create resistance and improve expiratory volume, and Segmental Breathing, which enhances inspiratory volume for lung expansion. In contrast, Incentive Spirometry provides visual feedback to guide deep inhalation; it includes both upside and upside-down usage of the spirometer for the maintenance of pulmonary function and preventing alveolar collapse.

Conducted as a randomized clinical trial, this study will include 40 pediatric participants aged 5-16, recruited from Gulab Devi Chest Hospital and Children's Hospital, Lahore. Participants will be randomly divided into two groups: one receiving Bubble PEP with Segmental Breathing and the other using Incentive Spirometry, both combined with conventional chest physiotherapy and mobility. Outcome measures, including lung expansion (via X-ray), dyspnea (assessed using the Pediatric Dyspnea Scale), chest expansion (measured with a measuring tape), oxygen saturation (SpO₂), and respiratory rate, will be recorded pre- and post-intervention. The study hypothesises that the Bubble PEP and Segmental Breathing approach may offer a cost-effective and efficient alternative to Incentive Spirometry, particularly for patients who cannot afford mechanical devices. Statistical analysis will be performed using SPSS version 2023 to determine the intervention's effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 to 16.
* Suffering from Pleural effusion or hydrothorax.
* Thoracic drainage system in situ for 24 hours.
* Either gender will be included.
* Patients without any other co-existing illness.

Exclusion Criteria:

* Any other pulmonary pathology that does not fit the diagnostic criteria of Pleural Effusion.
* Participants with unbearable chest pain, chylothorax, hemothorax, pneumothorax, chest trauma or rib fracture.
* Participants with other comorbidities leading to pleural effusion.
* Patients who have chest musculoskeletal deformities.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Lung Expansion | Baseline, 2 weeks
  To assess lung expansion before and after the intervention, anteroposterior chest X-rays will be used to evaluate improvements in lung volume and potential reductions in pleural effusion. This method allows for the measurement of lung field dimensions, changes in the opacity of lung areas affected by pleural effusion, and overall changes in thoracic structure that might indicate therapeutic effectiveness.
Pediatric Dyspnea Scale | Baseline, 2 weeks
  The Pediatric Dyspnea Scale (PDS) assesses subjective dyspnea in pediatric patients by using a visual and numerical scale, where patients indicate their perception of breathlessness. The PDS is scored from 1 through 7 where 1 indicates "No trouble at all" breathing and 7 indicates "Very much trouble" and a score of 1 through 7 was assigned accordingly.

SECONDARY OUTCOMES:
Chest Expansion | Baseline, 2 weeks
  Chest expansion will be measured with the help of tape method at different stages of the chest which measures symmetry and extent of expansion. The levels of measurements are at sternal notch, at xiphoid process and at T8vertebral level.
Oxygen Saturation | Baseline, 2 weeks
  Oxygen saturation (SpO2) will be measured using a pulse oximeter to evaluate improvements in oxygenation resulting from enhanced lung function.
Respiratory Rate | Baseline, 2 weeks
  The respiratory rate can be manually counted or evaluated using respiratory monitoring equipment, offering an objective measure of respiratory efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Tayyba Bari, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- The Children Hospital and University of Child Health Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dos Santos EDC, da Silva JS, de Assis Filho MTT, Vidal MB, Monte MC, Lunardi AC. Adding positive airway pressure to mobilisation and respiratory techniques hastens pleural drainage: a randomised trial. J Physiother. 2020 Jan;66(1):19-26. doi: 10.1016/j.jphys.2019.11.006. Epub 2019 Dec 13. PMID 31843426